CLINICAL TRIAL: NCT03158090
Title: The Longitudinal Approach to Acromegaly: A Pattern of Treatment and Comparative Effectiveness Research
Status: Recruiting | Type: Observational
Sponsor: Ginkgo Leaf Center for Rare Disorders (Other)
Responsible Party: Sponsor
Other Study IDs: Titan
Record Dates: First submitted 2017-05-06; First posted 2017-05-17 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Acromegaly
Keywords: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — Octreotide; lanreotide; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Surgical treatment: The subject was received transnasal butterfly surgery.
  Interventions: Procedure: Transnasal butterfly surgery
- Drug therapy: The subject was received drug treatment including somatostatin analogues such as sandostatin and lanreotide, dopamine receptor agonists and GH receptor antagonists.
  Interventions: Drug: sandostatin
- Radiotherapeutics: he subject was received radiotherapy methods including radiotherapy, linear accelerator X knife, gamma knife and so on.
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Procedure: Transnasal butterfly surgery — The patient will be treated in accordance with the advice of the local doctor in charge, and this study does not interfere with any treatment of the patient.
  Groups: Surgical treatment
Drug: sandostatin — The patient will be treated in accordance with the advice of the local doctor in charge, and this study does not interfere with any treatment of the patient
  Other Names: Lanreotide
  Groups: Drug therapy
Radiation: radiotherapy — The patient will be treated in accordance with the advice of the local doctor in charge, and this study does not interfere with any treatment of the patient
  Groups: Radiotherapeutics

SUMMARY:
This study is a prospective, noninteractive, observational, and longitudinal study aimed at assessing the treatment pattern and clinical outcome of acromegaly in China.

DETAILED DESCRIPTION:
The study was designed to answer some of the most important questions about the treatment modalities of acromegaly, the relevance of these treatment modalities to patients' clinical outcomes and the economic impact of treatment programs on patients. These answers may be of great help to the treatment of these populations and may also help to make treatment and related health decisions in the future.

This study only collects the patient's medical information during the study and does not interfere with the patient's treatment. Each patient will be assigned a unique patient identification number for the study. The sites will maintain a confidential decode list that enables the study staff at the site to link the assigned patient identification number with the patient's medical records for extraction of study-required data. These registries will be maintained following International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) and the respective local privacy laws and requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Be able and willing to sign the informed consent form (ICF)
2. Male, female, age 18-75 years old (including 18 years old and 75 years old).
3. Compliance with acromegaly diagnostic criteria:

   * At least one laboratory or medical record shows that the patient is random GH ≥ 2.5 μg / L
   * At least one checklist or medical record shows radiographic evidence that the patient has a pituitary tumor

Exclusion Criteria:

1. Ectopic secretion of GH or pituitary cancer
2. The patient is diagnosed with other complicated malignancies, or has previously been diagnosed with another malignancy, and there is currently evidence of lesion residue.
3. Have a diagnosis of other severe acute or chronic medical or psychiatric conditions that may increase the risk associated with study participation or may interfere with the interpretation of the study results and, in the judgement of the Investigator, would make the patient inappropriate for enrollment in this study.
4. Be a patient who, in the judgement of the Investigator, would be inappropriate for enrollment in this study

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chinese adult acromegaly patients are invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1965 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2050-12-30 (Estimated); Study Completion 2051-01-30 (Estimated)

PRIMARY OUTCOMES:
clinical outcome: overall survival | 30 yeas
  To compare overall survival of acromegaly in China between receiving surgery, drug and radiotherapeutics treatment

SECONDARY OUTCOMES:
clinical efficacy: control required GH level | 30 years
  To compare control required GH level of different treatment models (surgery, drug and radiotherapeutics treatment) in patients with acromegaly in China
Cost-effectiveness | 30 years
  To compare cost for acromegaly of different treatment models (surgery, drug and radiotherapeutics treatment) in patients with acromegaly in China

CONTACTS AND LOCATIONS:
Locations (1):
- China Acromegaly Organization, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided